CLINICAL TRIAL: NCT03157128
Title: A Phase 1/2 Study of Oral Selpercatinib (LOXO-292) in Patients With Advanced Solid Tumors, Including RET Fusion-Positive Solid Tumors, Medullary Thyroid Cancer, and Other Tumors With RET Activation (LIBRETTO-001)
Brief Title: A Study of Selpercatinib (LOXO-292) in Participants With Advanced Solid Tumors, RET Fusion-Positive Solid Tumors, and Medullary Thyroid Cancer (LIBRETTO-001)
Acronym: LIBRETTO-001
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17477; J2G-OX-JZJA (Other: Eli Lilly and Company); LOXO-RET-17001 (Other: Loxo Oncology, Inc.); 2017-000800-59 (EudraCT Number)
Expanded Access: NCT03906331 (Approved for marketing)
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer; Medullary Thyroid Cancer; Colon Cancer; Any Solid Tumor
Keywords: LOXO-292; KIF5B-RET; M918T; CCDC6-RET; RET-PTC1; NCOA4-RET; RET-PTC; RET-PTC3; RET-PTC4; PRKAR1A-RET; RET-PTC2; GOLGA5-RET; RET-PTC5; ERC1-RET; KTN1-RET; RET-PTC8; HOOK3-RET; PCM1-RET; TRIM24-RET; RET-PTC6; TRIM27-RET; TRIM33-RET; RET-PTC7; AKAP13-RET; FKBP15-RET; SPECC1L-RET; TBL1XR1-RET; BCR-RET; FGRF1OP-RET; RFG8-RET; RET-PTC9; ACBD5-RET; MYH13-RET; CUX1-RET; KIAA1468-RET; FRMD4A-RET; SQSTM1-RET; AFAP1L2-RET; PPFIBP2-RET; EML4-RET; PARD3-RET; G533C; C609F; C609G; C609R; C609S; C609Y; C611F; C611G; C611S; C611Y; C611W; C618F; C618R; C618S; C620F; C620R; C620S; C630R; C630Y; D631Y; C634F; C634G; C634R; C634S; C634W; C634Y; K666E; E768D; L790F; V804L; V804M; A883F; S891A; R912P; CLIP1-RET; Y806C; RET fusion; RET alteration; RET mutation; RET rearrangement; RET translocation; Neoplasms by Site; Neoplasms; Non-Small Cell Lung Cancer; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Respiratory Tract Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Medullary Thyroid Cancer; Papillary Thyroid Cancer; Thyroid Diseases; Thyroid Neoplasms; Cancer of the Thyroid; Cancer of Thyroid; Neoplasms, Thyroid; Thyroid Ademona; Thyroid Cancer; Thyroid Carcinoma; Endocrine System Diseases; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Thoracic Neoplasms; CNS tumor; Primary CNS tumor; Cancer of Colon; Cancer of the Colon; Colon Cancer; Colon Neoplasms; Colonic Cancer; Neoplasms, Colonic; Malignant tumor of Breast; Mammary Cancer; Mammary Carcinoma, Human; Mammary Neoplasm, Human; Neoplasms, Breast; Tumors, Breast; Human Mammary Carcinoma; Malignant Neoplasm of Breast; Breast Carcinoma; Breast Tumors; Cancer of the Breast; Breast Neoplasms; Breast Cancer; RET Inhibitor; MTC; NSCLC; selpercatinib; neo-adjuvant treatment in early stage NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Medullary; Colonic Neoplasms; Neoplasms by Site; Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Thyroid Cancer, Papillary; Thyroid Diseases; Thyroid Neoplasms; Endocrine System Diseases; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Thoracic Neoplasms; Central Nervous System Neoplasms; Breast Neoplasms | interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LOXO-292 (Experimental): Phase 1 - Multiple doses of LOXO-292 (selpercatinib) Phase 2 - The maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D)
  Interventions: Drug: LOXO-292

INTERVENTIONS:
Drug: LOXO-292 — Oral LOXO-292
  Other Names: Selpercatinib; LY3527723

SUMMARY:
This is an open-label, first-in-human study designed to evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary anti-tumor activity of selpercatinib (also known as LOXO-292) administered orally to participants with advanced solid tumors, including rearranged during transfection (RET)-fusion-positive solid tumors, medullary thyroid cancer (MTC) and other tumors with RET activation.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase 1/2 study in participants with advanced solid tumors, including RET fusion-positive solid tumors, MTC, and other tumors with RET activation. The trial will be conducted in 2 parts: Phase 1 (dose escalation - completed) and phase 2 (dose expansion). Participants with advanced cancer are eligible if they have progressed on or are intolerant to available standard therapies, or no standard or available curative therapy exists, or in the opinion of the Investigator, they would be unlikely to tolerate or derive significant clinical benefit from appropriate standard of care therapy, or they declined standard therapy. A dose of 160 milligrams (mg) twice a day (BID) has been selected as the recommended phase 2 dose (RP2D). Approximately 875 participants with advanced solid tumors harboring a RET gene alteration in tumor and/or blood will be enrolled to one of seven phase 2 cohorts:

* Cohort 1: Advanced RET fusion positive solid tumor other than NSCLC or thyroid cancer for participants who progressed on or intolerant to first line therapy (open)
* Cohort 2: Advanced RET fusion positive solid tumor other than NSCLC or thyroid cancer for treatment naïve participants (open)
* Cohort 3: Advanced RET-mutant MTC participants who progressed on or intolerant to first line therapy (closed)
* Cohort 4: Advanced RET-mutant MTC participants who are treatment naïve (closed)
* Cohort 5: Advanced RET-altered solid tumor for participants other than NSCLC or thyroid cancer and RET-mutant MEN2 spectrum tumors (e.g. pheochromocytoma) otherwise ineligible for cohorts 1-4. See details in inclusion/exclusion criteria (open)
* Cohort 6: Participants otherwise eligible for Cohorts 1-5 who discontinued another RET inhibitor due to intolerance may be eligible with prior Sponsor approval (closed)
* Cohort 7: RET fusion positive early-stage non-small cell lung cancer (NSCLC) participants who are candidates for definitive surgery. Participants will receive selpercatinib in a neoadjuvant and adjuvant setting. Participants will be followed for disease recurrence for up to 5 years from the date of surgery (closed)

ELIGIBILITY:
Key Inclusion Criteria:

For Phase 1:

* Participants with a locally advanced or metastatic solid tumor that:
* Has progressed on or is intolerant to standard therapy, or
* For which no standard therapy exists, or in the opinion of the Investigator, are not candidates for or would be unlikely to tolerate or derive significant clinical benefit from standard therapy, or
* Decline standard therapy
* Prior multikinase inhibitors (MKIs) with anti-RET activity are allowed
* A RET gene alteration is not required initially. Once adequate PK exposure is achieved, evidence of RET gene alteration in tumor and/or blood is required as identified through molecular assays, as performed for clinical evaluation
* Measurable or non-measurable disease as determined by RECIST 1.1 or RANO as appropriate to tumor type
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2 or Lansky Performance Score (LPS) greater than or equal to (≥) 40 percent (%) (age less than [<] 16 years) with no sudden deterioration 2 weeks prior to the first dose of study treatment
* Adequate hematologic, hepatic and renal function
* Life expectancy of at least 3 months

For Phase 2: As for phase 1 with the following modifications:

* For Cohort 1: Participants must have received prior standard therapy appropriate for their tumor type and stage of disease, or in the opinion of the Investigator, would be unlikely to tolerate or derive clinical benefit from appropriate standard of care therapy
* Cohorts 1 and 2:

  * Enrollment will be restricted to participants with evidence of a RET gene alteration in tumor
  * At least one measurable lesion as defined by RECIST 1.1 or RANO, as appropriate to tumor type and not previously irradiated
* Cohorts 3 and 4: Enrollment closed
* Cohort 5:

  * Cohorts 1-4 without measurable disease
  * MCT not meeting the requirements for Cohorts 3 or 4
  * MTC syndrome spectrum cancers (e.g., MTC, pheochromocytoma), cancers with neuroendocrine features/differentiation, or poorly differentiated thyroid cancers with other RET alteration/activation may be allowed with prior Sponsor approval
  * cfDNA positive for a RET gene alteration not known to be present in a tumor sample
* Cohort 6: Participants who otherwise are eligible for Cohorts 1, 2 or 5 who discontinued another RET inhibitor may be eligible with prior Sponsor approval
* Cohort 7: Participants with a histologically confirmed stage IB-IIIA NSCLC and a RET fusion; determined to be medically operable and tumor deemed resectable by a thoracic surgical oncologist, without prior systemic treatment for NSCLC

Key Exclusion Criteria (Phase 1 and Phase 2):

* Phase 2 Cohorts 1 and 2: an additional known oncogenic driver
* Cohorts 3 and 4: Enrollment closed
* Cohorts 1, 2 and 5: prior treatment with a selective RET inhibitor Notes: Participants otherwise eligible for Cohorts 1, 2, and 5 who discontinued another selective RET inhibitor may be eligible for Phase 2 Cohort 6 with prior Sponsor approval
* Investigational agent or anticancer therapy (including chemotherapy, biologic therapy, immunotherapy, anticancer Chinese medicine or other anticancer herbal remedy) within 5 half-lives or 2 weeks (whichever is shorter) prior to planned start of LOXO-292 (selpercatinib). In addition, no concurrent investigational anti-cancer therapy is permitted Note: Potential exception for this exclusion criterion will require a valid scientific justification and approval from the Sponsor
* Major surgery (excluding placement of vascular access) within 2 weeks prior to planned start of LOXO-292 (selpercatinib)
* Radiotherapy with a limited field of radiation for palliation within 1 week of planned start of LOXO-292 (selpercatinib), with the exception of participants receiving radiation to more than 30% of the bone marrow or with a wide field of radiation, which must be completed at least 4 weeks prior to the first dose of study treatment
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy
* Symptomatic primary CNS tumor, metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression. Participants are eligible if neurological symptoms and CNS imaging are stable and steroid dose is stable for 14 days prior to the first dose of LOXO-292 (selpercatinib) and no CNS surgery or radiation has been performed for 28 days, 14 days if stereotactic radiosurgery (SRS)
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to planned start of LOXO-292 (selpercatinib) or prolongation of the QT interval corrected (QTcF) greater than (>) 470 milliseconds (msec)

  * Participants with implanted pacemakers may enter the study without meeting QTc criteria due to nonevaluable measurement if it is possible to monitor for QT changes.
  * Participants with bundle branch block may be considered for study entry if QTc is appropriate by a formula other than Fridericia's and if it is possible to monitor for QT changes.
* Required treatment with certain strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and certain prohibited concomitant medications
* Phase 2 Cohort 7 (neoadjuvant treatment): Participant must not have received prior systemic therapy for NSCLC.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1: MTD | The first 28 days of treatment (Cycle 1)
  Incidence rate and category of dose limiting toxicities (DLTs) during the first 28-day cycle of LOXO-292 (selpercatinib) treatment
Phase 1: RP2D | The first 28 days of treatment (Cycle 1) and every cycle (28 days) for approximately 12 months (or earlier if the participant discontinues from the study)
  Phase 1: RP2D
Phase 2: Objective Response Rate | Approximately every 8 weeks for one year, then every 12 weeks, and 7 days after the last dose (for up to 2 years) in participants who have not progressed.
  As assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Response Assessment in Neuro-Oncology (RANO), as appropriate to tumor type, as assessed by independent review committee (IRC)

SECONDARY OUTCOMES:
Phase 1: Number of Participants with a Treatment-Related Adverse Event(s) (TRAE[s]) | From the time of informed consent, for approximately 24 months (or earlier if the participant discontinues from the study), and through Safety Follow-up (28 days after the last dose)
  Phase 1: Number of Participants with a TRAE(s)
Phase 1: Number of Participants with an Abnormal Laboratory or Physical Exam Result(s) | From the time of informed consent, for approximately 24 months (or earlier if the participant discontinues from the study), and through Safety Follow-up (28 days after the last dose)
  Phase 1: Number of Participants with an Abnormal Laboratory or Physical Exam Result(s)
Phase 1: Overall Response Rate (ORR) based on RECIST 1.1 or RANO, as Appropriate to Tumor Type | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 1: ORR based on RECIST 1.1 or RANO, as Appropriate to Tumor Type
Phase 2: ORR (by Investigator) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: ORR (by Investigator)
Phase 2: Best Change in Tumor Size from Baseline (by IRC and Investigator) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: Best Change in Tumor Size from Baseline (by IRC and Investigator)
Phase 2: Duration of Response (DOR; by IRC and Investigator) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: DOR (by IRC and Investigator)
Phase 2: Central Nervous System (CNS) ORR (by IRC) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: CNS ORR (by IRC)
Phase 2: CNS DOR (by IRC) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: CNS DOR (by IRC)
Phase 2: Time to Any and Best Response (by IRC and Investigator) | every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: Time to Any and Best Response (by IRC and Investigator)
Phase 2: CBR (by IRC and Investigator) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: CBR (by IRC and Investigator)
Phase 2: PFS (by IRC and Investigator) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: PFS (by IRC and Investigator)
Phase 2: Overall Survival (OS) | Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed
  Phase 2: OS
Phase 2: Percentage of Participants with any Serious Adverse Event (SAE[s]) | From the time of informed consent, for approximately 24 months (or earlier if the participant discontinues from the study), and through Safety Follow-up (28 days after the last dose)
  Phase 2: Percentage of Participants with any SAE(s)
Phase 1 and 2: Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve of LOXO-292 (Selpercatinib) | Cycle 1 Day 1 through Cycle 5 Day 1 (Cycle = 28 days)
  Phase 1 and 2: PK: AUC of LOXO-292 (Selpercatinib)
Phase 1 and 2: PK: Maximum Concentration (Cmax) of LOXO-292 (Selpercatinib) | Cycle 1 Day 1 through Cycle 5 Day 1 (Cycle = 28 days)
  Phase 1 and 2: PK: Cmax of LOXO-292 (Selpercatinib)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (85):
- United States (41):
  - Mayo Clinic of Scottsdale, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente, Oakland, California
  - Irvine Medical Center, Orange, California
  - University of California - San Diego, San Diego, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Kaiser Permanente Medical Center, Walnut Creek, California
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Memorial Hospital Pembroke, Pembroke, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago Medicine-Comprehensive Cancer Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - USO-Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- BC Cancer Vancouver, Vancouver, British Columbia, Canada
- Rigshospitalet, Copenhagen, Denmark
- France (6):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - APHM Hôpital de la Timone, Marseille
  - Institut du Cancer de Montpellier - Val d'aurelle, Montpellier
  - Gustave Roussy, Villejuif
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
- Prince of Wales Hospital, Hong Kong, Shatin, New Territories, Hong Kong
- Israel (4):
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center - Pediatric Outpatient Clinic, Beersheba
  - Hadassah Medical Center, Jerusalem
- Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- Japan (13):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kindai University Hospital, Osaka Sayama-shi, Osaka
  - Tominaga Hospital, Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
- National Cancer Centre Singapore, Singapore, Central Singapore, Singapore
- South Korea (5):
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gautschi O, Park K, Solomon BJ, Tomasini P, Loong HH, De Braud F, Goto K, Peterson P, Barker S, Liming K, Oxnard GR, Frimodt-Moller B, Drilon A. Selpercatinib in RET Fusion-Positive Non-Small Cell Lung Cancer: Final Safety and Efficacy, Including Overall Survival, From the LIBRETTO-001 Phase I/II Trial. J Clin Oncol. 2025 May 20;43(15):1758-1764. doi: 10.1200/JCO-24-02076. Epub 2025 Feb 21. PMID 39983053
- [Derived] Wirth LJ, Brose MS, Subbiah V, Worden F, Solomon B, Robinson B, Hadoux J, Tomasini P, Weiler D, Deschler-Baier B, Tan DSW, Maeda P, Lin Y, Singh R, Bayt T, Drilon A, Cassier PA. Durability of Response With Selpercatinib in Patients With RET-Activated Thyroid Cancer: Long-Term Safety and Efficacy From LIBRETTO-001. J Clin Oncol. 2024 Sep 20;42(27):3187-3195. doi: 10.1200/JCO.23.02503. Epub 2024 Aug 2. PMID 39094065
- [Derived] Deschler-Baier B, Krebs M, Kroiss M, Chatterjee M, Gundel D, Kestler C, Kerscher A, Kunzmann V, Appenzeller S, Maurus K, Rosenwald A, Bargou R, Gerhard-Hartmann E, Venkataramani V. Rapid response to selpercatinib in RET fusion positive pancreatic neuroendocrine carcinoma confirmed by smartwatch. NPJ Precis Oncol. 2024 Jul 31;8(1):167. doi: 10.1038/s41698-024-00659-x. PMID 39085487
- [Derived] Deschler-Baier B, Konda B, Massarelli E, Hu MI, Wirth LJ, Xu X, Wright J, Clifton-Bligh RJ. Clinical Activity of Selpercatinib in RET-mutant Pheochromocytoma. J Clin Endocrinol Metab. 2025 Feb 18;110(3):e600-e606. doi: 10.1210/clinem/dgae283. PMID 38661071
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Duke ES, Bradford D, Marcovitz M, Amatya AK, Mishra-Kalyani PS, Nguyen E, Price LSL, Fourie Zirkelbach J, Li Y, Bi Y, Kraft J, Dorff SE, Scepura B, Stephenson M, Ojofeitimi I, Nair A, Han Y, Tezak Z, Lemery SJ, Pazdur R, Larkins E, Singh H. FDA Approval Summary: Selpercatinib for the Treatment of Advanced RET Fusion-Positive Solid Tumors. Clin Cancer Res. 2023 Sep 15;29(18):3573-3578. doi: 10.1158/1078-0432.CCR-23-0459. PMID 37265412
- [Derived] Murciano-Goroff YR, Falcon CJ, Lin ST, Chacko C, Grimaldi G, Liu D, Wilhelm C, Iasonos A, Drilon A. Central Nervous System Disease in Patients With RET Fusion-Positive NSCLC Treated With Selpercatinib. J Thorac Oncol. 2023 May;18(5):620-627. doi: 10.1016/j.jtho.2023.01.008. Epub 2023 Jan 16. PMID 36657661
- [Derived] Drilon A, Subbiah V, Gautschi O, Tomasini P, de Braud F, Solomon BJ, Shao-Weng Tan D, Alonso G, Wolf J, Park K, Goto K, Soldatenkova V, Szymczak S, Barker SS, Puri T, Bence Lin A, Loong H, Besse B. Selpercatinib in Patients With RET Fusion-Positive Non-Small-Cell Lung Cancer: Updated Safety and Efficacy From the Registrational LIBRETTO-001 Phase I/II Trial. J Clin Oncol. 2023 Jan 10;41(2):385-394. doi: 10.1200/JCO.22.00393. Epub 2022 Sep 19. PMID 36122315
- [Derived] Subbiah V, Wolf J, Konda B, Kang H, Spira A, Weiss J, Takeda M, Ohe Y, Khan S, Ohashi K, Soldatenkova V, Szymczak S, Sullivan L, Wright J, Drilon A. Tumour-agnostic efficacy and safety of selpercatinib in patients with RET fusion-positive solid tumours other than lung or thyroid tumours (LIBRETTO-001): a phase 1/2, open-label, basket trial. Lancet Oncol. 2022 Oct;23(10):1261-1273. doi: 10.1016/S1470-2045(22)00541-1. Epub 2022 Sep 12. PMID 36108661
- [Derived] Rolfo C, Hess LM, Jen MH, Peterson P, Li X, Liu H, Lai Y, Sugihara T, Kiiskinen U, Vickers A, Summers Y. External control cohorts for the single-arm LIBRETTO-001 trial of selpercatinib in RET+ non-small-cell lung cancer. ESMO Open. 2022 Aug;7(4):100551. doi: 10.1016/j.esmoop.2022.100551. Epub 2022 Aug 2. PMID 35930972
- [Derived] Subbiah V, Gainor JF, Oxnard GR, Tan DSW, Owen DH, Cho BC, Loong HH, McCoach CE, Weiss J, Kim YJ, Bazhenova L, Park K, Daga H, Besse B, Gautschi O, Rolfo C, Zhu EY, Kherani JF, Huang X, Kang S, Drilon A. Intracranial Efficacy of Selpercatinib in RET Fusion-Positive Non-Small Cell Lung Cancers on the LIBRETTO-001 Trial. Clin Cancer Res. 2021 Aug 1;27(15):4160-4167. doi: 10.1158/1078-0432.CCR-21-0800. Epub 2021 Jun 4. PMID 34088726
- [Derived] Wirth LJ, Sherman E, Robinson B, Solomon B, Kang H, Lorch J, Worden F, Brose M, Patel J, Leboulleux S, Godbert Y, Barlesi F, Morris JC, Owonikoko TK, Tan DSW, Gautschi O, Weiss J, de la Fouchardiere C, Burkard ME, Laskin J, Taylor MH, Kroiss M, Medioni J, Goldman JW, Bauer TM, Levy B, Zhu VW, Lakhani N, Moreno V, Ebata K, Nguyen M, Heirich D, Zhu EY, Huang X, Yang L, Kherani J, Rothenberg SM, Drilon A, Subbiah V, Shah MH, Cabanillas ME. Efficacy of Selpercatinib in RET-Altered Thyroid Cancers. N Engl J Med. 2020 Aug 27;383(9):825-835. doi: 10.1056/NEJMoa2005651. PMID 32846061
- [Derived] Drilon A, Oxnard GR, Tan DSW, Loong HHF, Johnson M, Gainor J, McCoach CE, Gautschi O, Besse B, Cho BC, Peled N, Weiss J, Kim YJ, Ohe Y, Nishio M, Park K, Patel J, Seto T, Sakamoto T, Rosen E, Shah MH, Barlesi F, Cassier PA, Bazhenova L, De Braud F, Garralda E, Velcheti V, Satouchi M, Ohashi K, Pennell NA, Reckamp KL, Dy GK, Wolf J, Solomon B, Falchook G, Ebata K, Nguyen M, Nair B, Zhu EY, Yang L, Huang X, Olek E, Rothenberg SM, Goto K, Subbiah V. Efficacy of Selpercatinib in RET Fusion-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Aug 27;383(9):813-824. doi: 10.1056/NEJMoa2005653. PMID 32846060